CLINICAL TRIAL: NCT03862248
Title: Novel Triple-dose Tuberculosis Retreatment Regimens: How to Overcome Resistance Without Creating More
Acronym: TriDoRe
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Feasibility of the clinical trial could not be confirmed at the different sites.
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Damien Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TriDoRe
Record Dates: First submitted 2019-02-04; First posted 2019-03-05 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Dose Isoniazid (Experimental): New high-dose isoniazid retreatment regimen (6EH³RZ) - H 15mg/kg
  Interventions: Drug: 6EH³RZ
- High-Dose Rifampicin (Experimental): New high-dose rifampicin retreatment regimen (6EHR³Z) - R 30mg/kg
  Interventions: Drug: 6EHR³Z
- World Health Organisation (WHO) regimen (Active Comparator): WHO levofloxacin-strengthened regimen (6EHRZLfx)
  Interventions: Drug: 6EHRZLfx

INTERVENTIONS:
Drug: 6EH³RZ — New high-dose isoniazid retreatment regimen (6EH³RZ) - H 15mg/kg
  Arms: High-Dose Isoniazid
Drug: 6EHR³Z — New high-dose rifampicin retreatment regimen (6EHR³Z) - R 30mg/kg
  Arms: High-Dose Rifampicin
Drug: 6EHRZLfx — WHO levofloxacin-strengthened regimen (6EHRZLfx)
  Arms: World Health Organisation (WHO) regimen

SUMMARY:
Drug-resistance is a major challenge for tuberculosis (TB) care programs. The new WHO guideline recommends adding levofloxacin in previously treated patients with isoniazid-resistant rifampicin-susceptible TB. The investigators believe that such a retreatment regimen may result in acquired resistance to fluoroquinolone, the core drug of multidrug-resistant TB (MDR-TB) regimen, and thus threaten the effectiveness of the fluoroquinolone-based MDR-TB treatment regimen. Therefore the investigators propose to study if regimens strengthened by using high-dose first-line drugs, either a triple dose of isoniazid or a triple dose of rifampicin, are non-inferior to the WHO recommended levofloxacin-strengthened regimen. If one of both high-dose regimens would be non-inferior, it could replace the levofloxacin-strengthened regimen.

ELIGIBILITY:
Inclusion Criteria:

* All newly registered patients with smear-positive recurrent pulmonary TB
* Adults as well as children (no age limit)
* Able and willing to provide written informed consent

Exclusion Criteria:

* Patients transferred to a health facility not supported by Damien Foundation will be excluded. This includes patients diagnosed with HIV/TB-coinfection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity
Enrollment: 0 (Actual)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Bacteriological effectiveness (proportion of relapse-free cure excluding deaths and lost-to-follow-up) | 18 months (6-month treatment + 12-month follow-up period)
  To study if the bacteriological effectiveness of two high-dose regimens is non-inferior to the WHO recommended levofloxacin-strengthened regimen in patients with rifampicin-susceptible recurrent TB. Relapse-free cure is based on sputum smear and culture-result.

SECONDARY OUTCOMES:
Frequency of resistance to the different drug components at screening. | At screening (day 0)
  Determine the initial resistance profile to the different drug components (Isoniazid, Rifampicin, Pyrazinamide and Levofloxacin) for the entire cohort of patients with recurrent TB
Identify predictors of bacteriological effectiveness | 18 months (6-month treatment + 12-month follow-up period)
  Identify predictors (including treatment regimen, resistance profile, presence of cavities, the grading of the smear, …) of bacteriological effectiveness
Programmatic effectiveness (i.e proportion of participants with relapse-free cure) | 18 months (6-month treatment + 12-month follow-up period)
  Compare the programmatic effectiveness of the 3 different regimens. Relapse-free cure is based on sputum smear and culture-result.
Number of SAEs and study-specific adverse events of the different retreatment regimens | up to month 6
  Compare the safety (SAEs and study-specific adverse events ) of the different retreatment regimens.
Negative predictive value of two-week FDA | 2 weeks after start of treatment
  Evaluate a novel application of fluorescein diacetate vital staining fluorescence microscopy (FDA) at 0 and 2 weeks of treatment, to estimate its utility as screening test for initial resistance to rifampicin, and identify predictors for FDA reduction at 2 weeks. The negative predictive value of two-week FDA showing no lack of 10-fold reduction of viable bacilli at two weeks.
Proportion of participants relapse-free cure | 18 months (6-month treatment + 12-month follow-up period)
  To estimate the proportion of relapse-free cure among patients with FDA conversion to zero at 2 weeks, by regimen.The proportion (95% confidence interval) relapse-free cure among those who converted on the two-week FDA, by regimen.
Difference (95% confidence interval) in bacteriological effectiveness (susceptible to both rifampicin and isoniazid vs heteroresistance to rifampicin and/or isoniazid).(heteroresistance), by regimen studied in the trial | 18 months (6-month treatment + 12-month follow-up period)
  Estimate the clinical relevance of different proportions of mutant subpopulations (heteroresistance), by regimen studied in the trial.
Proportion of participants with acquired resistance | 18 months (6-month treatment + 12-month follow-up period)
  proportion of participants with acquired resistance, by treatment regimen
Identify predictors of programmatic effectiveness (including treatment regimen, resistance profile, presence of cavities, the grading of the smear, …) | 18 months (6-month treatment + 12-month follow-up period)
  Identify predictors (including treatment regimen, resistance profile, presence of cavities, the grading of the smear, …).

CONTACTS AND LOCATIONS:
Overall Officials: Tom Decroo, MD, Principal Investigator — Insitute of Tropical Medicine Antwerp
Locations (1):
- Damien Foundation, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No